CLINICAL TRIAL: NCT04102202
Title: A Phase IIa, Randomized, Double-Blind, Placebo-Controlled, Parallel-Groups, Safety & Efficacy Trial of BOL-DP-o-05 as an Add-On Treatment for Preservation of Beta-Cell Function in Subjects With Newly-Diagnosed T1DM
Brief Title: BOL-DP-o-05 as an Add-On Treatment of Subjects With Newly Diagnosed Type 1 Diabetes Mellitus
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to company strategic decision
Sponsor: Breath of Life International Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BOL-P-023
Record Dates: First submitted 2019-09-15; First posted 2019-09-25 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Type1 Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BOL-DP-o-05 (Experimental)
  Interventions: Drug: BOL-DP-o-05
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BOL-DP-o-05 — BOL-DP-o-05
  Arms: BOL-DP-o-05
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
BOL-DP-o-05 as an Add-On Treatment for Preservation of Beta-Cell Function in Subjects With Newly-Diagnosed Type 1 Diabetes Mellitus (T1DM)

DETAILED DESCRIPTION:
A Randomized, Double-Blind, Placebo-Controlled, Parallel-Groups study in which subjects will be randomized to receive either BOL-DP-o-05 or placebo as an Add-On Treatment. The study evaluates the effect of BOL-DP-o-05 for Preservation of Beta-Cell Function in Subjects with Newly-Diagnosed Type 1 Diabetes Mellitus (T1DM). The study includes a screening period up to three weeks followed by a 48-week treatment period

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities.
* T1DM ≤ 20 weeks prior to screening.
* Male or female, aged 5-30 years old (both inclusive) at the time of signing the informed consent form.
* Non-fasting peak C-peptide ≥0.2 nmol/l during mixed-meal tolerance test (MMTT) at Visit 1.
* BMI ≥18.5 kg/m2.
* Presence of one or more islet-specific autoantibodies at the screening.
* Insulin dependence, unless in temporary spontaneous remission ("honeymoon period").

Exclusion Criteria:

* Daily insulin usage > 1 U/kg per day at screening
* History of recurrent (e.g. several times a year) of severe (e.g. pneumonia) or chronic infections or conditions predisposing to chronic infections.
* History of severe systemic fungal infection within the past 12 months prior to screening unless treated and resolved with appropriate documented therapy.
* Vaccination within 4 weeks before randomization.
* Receipt of any other concomitant medications or herbal products that can influence the immune system within 90 days prior to screening.
* History of pancreatitis (acute or chronic).
* Any past or current diagnosis of malignant neoplasms.
* Known impairment of the immune system, except for T1DM, coeliac disease, alopecia, autoimmune antibodies not considered clinical important (e.g. thyroid antibodies without any clinically important thyroid disease), and vitiligo.
* Patients with a psychiatric condition (e.g. severe anxiety, psychosis) that would interfere with the study as determined by the primary investigator.
* Patients with known allergy to one or more of the study drug components.
* Female patients who are pregnant, lactating, or who want to get pregnant during the study period. In the case of young patients, the PI should raise this point with the patient/family.
* Male subjects who want their partner to get pregnant.
* Female of child-bearing potential who do not agree to utilize medically acceptable and reliable means of birth control during the study and for 1 month following the last dose of the study unless the patient is young and the PI speaks with the patient/family and waived the criteria due to young age.
* Patients with a history of alcohol or any psychoactive substance abuse or dependence (including alcohol but excluding nicotine and caffeine).
* Patients with a first-degree family history of a psychiatric condition diagnosed at age<30 years.
* Patients with congestive heart failure or any other chronic disease.
* Patients with heart failure, psychotic state in the past, anxiety disorder, and heredity significant psychiatric inheritance in first-degree family relative, especially in patients younger than 30, and a history of addiction or drug abuse.

Ages: 5 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11-15 (Estimated); Primary Completion 2021-03-22 (Estimated); Study Completion 2021-03-22 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of BOL-DP-o-05 on preservation of beta-cell function | up to week 48
  Plasma levels of C-peptide concentration

SECONDARY OUTCOMES:
Number of diabetic ketoacidosis episodes | Through study completion, an average of 48 weeks
  Urine and plasma levels for ketones
Number of severe hypoglycaemic episodes | Through study completion, an average of 48 weeks
  Plasma glucose level
Peak MMTT stimulated C-peptide concentration | Base line and week 48
  Plasma levels of C-peptide concentration
To assess the change in fasting C-peptide | Baseline to week 24 and week 48
  Plasma levels of C-peptide concentration
To assess the change in HbA1c | Baseline to weeks 24 and 48
  HbA1c in plasma
To evaluate total daily insulin dose | Week 24 and week 48
  Insulin levels in units per kg
To Assess the percentage of patients that maintain stimulated peak C-peptide ≥ 0.2nmol/L | At week 48
  Plasma levels of C-peptide
To Assess the percentage of patients that achieve glycemic target of HbA1c ≤ 7.5% | At week 24 and week 48
  HbA1c in plasma
To assess the percent of subjects who require a daily insulin dose < 0.5 IU/kg body weight | After 12 months of first treatment
  Plasma glucose levels

IPD SHARING:
Plan to Share IPD: No